CLINICAL TRIAL: NCT01365377
Title: Impact of the Deliverance and Use of a Written Detailed Information Brochure on Anxiety Felt by the Family Members of Patients Admitted in Intensive Care Unit
Brief Title: Impact of Information Strategy Based on Booklet on Anxiety in Family in ICU
Acronym: FAMILLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Jean-Jacques ROUBY, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: FAMILLE-JJR-2
Record Dates: First submitted 2011-05-31; First posted 2011-06-03 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-04

CONDITIONS: Anxiety; Depression; Post-traumatic Stress Disorders
Keywords: Anxiety; Depression; Post-traumatic stress disorders; Quality of life; Family; ICU
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Booklet (Experimental): Referent member of the family is designated to receive a written detailed information on Critical care.
  Interventions: Other: booklet deliverance and use in the process of daily information
- No booklet (No Intervention): daily information to the family is given as usual.

INTERVENTIONS:
Other: booklet deliverance and use in the process of daily information — The brochure shows with text and pictures the day-living of the ICU ; Medical and para-medical staff and organization, the devices, complications and treatment
  Other Names: Brochure
  Arms: Booklet

SUMMARY:
Anxiety and depression are symptoms frequently met in ICU patients and relatives. Risk factors are known: disease severity, age, gender. Another risk factor is lack of information from the medical staff and nurses.

Anxiety and depression can be measured by the Hospital Anxiety and Depression Scale (HADS). Other scales are used in the psychiatric field : the Impact Event Score - Revisited (IES-R) is relevant to detect Post-Traumatic Stress Disorder (PTSD), The Short Form Health Survey (SF-36) is an assessment of life quality.

In the following study, the investigators will evaluate the impact of a "brochure" as complement of oral information on Anxiety developed by relatives and family of ICU patients.

The medical and surgical ICU is composed by two different units (different medical and nurse team, different location in the same hospital) of 12 beds on one side, 14 beds on the other side.

During a year, in the first unit, the investigators will use the booklet as support and complement of oral information : "booklet arm". The information process will be as usual in the other unit : "control arm". During the second year, the booklet will be used in the second unit while the first unit will return to the usual oral information (cross-over).

For each included patient, one relative or family member is pointed to be the referring family member or "referent". This "referent" receives the HADS questionnaire at Day 3 after admission, at day of discharge if the patient is alive, at one month after discharge. The IES-R questionnaire is delivered at discharge of the living patient and at day 30. The SF-36 questionnaire is given to the "referent" and the living patient at day 30. The day 30 questionnaires are send by mail at the "referent" address.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in ICU whose previsible length of stay is over 3 days.

Exclusion Criteria:

* Admitted patient without organ failure
* Family member or patient who can't speak and/or read French
* Family who didn't show off within the first week of hospitalization

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Decreased of the Anxiety Score of 20% in the "brochure arm" from admission to discharge of ICU. | One year per arm
  We hope to see the anxiety score decreasing between day of admission and day of discharge in the patient's relative who received the brocure.

SECONDARY OUTCOMES:
Decreased of Depression Scoring on the HADS | two years
  We hope to see a decreasing of the Depression Score, which is part of the Hospital Anxiety and Depression Scale, in the group of patient's relatives receiving the booklet.
Diagnostic and following of Post-traumatic stress disorder | Two years
  We hope to see a decreasing of the score in the Impact Event Score (Revisited)in the group of patient's relatives receiving the booklet, showing a less risk of PTSD.
Assessment of quality of life in patients and relatives | Two years
  A month after ICU discharge, we use the Short-Form 36 to assess quality of life of the surviving patients and their relative.

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit, Groupe Hospitalier Pitie-Salpetriere, Paris, France

REFERENCES:
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Jackson JC, Hart RP, Gordon SM, Shintani A, Truman B, May L, Ely EW. Six-month neuropsychological outcome of medical intensive care unit patients. Crit Care Med. 2003 Apr;31(4):1226-34. doi: 10.1097/01.CCM.0000059996.30263.94. PMID 12682497